CLINICAL TRIAL: NCT07098325
Title: Evaluation of Biological Reaction of Direct Three Dimensional Printed Retainers
Brief Title: Biological Reaction of Direct 3d Printed Retainers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Norhan Ibrahim Eldsokee Khidr, Principal Investigator, Master's Candidate at Orthodontic department at Al-Azhar University, Assiut branch., Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Direct 3d printed retainers
Record Dates: First submitted 2025-07-08; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Orthodontic Retainers
Keywords: Different thicknesses; Direct three dimensional printed retainers; Bacterial growth; Color change
MeSH Terms: interventions — Orthodontic Retainers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct 3d printed retainer of .5mm (Experimental): group wearing direct 3d retainer of .5 mm
  Interventions: Device: retainer with .5 mm thickness
- direct 3d printed retainer of 1mm (Experimental): group wearing direct 3 d retainer with thickness 1 mm
  Interventions: Device: retainer with 1 mm thickness

INTERVENTIONS:
Device: retainer with .5 mm thickness — direct 3d printed retainer with .5 mm thickness
  Arms: direct 3d printed retainer of .5mm
Device: retainer with 1 mm thickness — direct 3d printed retainer with 1 mm thickness,
  Arms: direct 3d printed retainer of 1mm

SUMMARY:
The aim of this study will be to evaluate the biological reaction of direct three dimensional printed retainers.

Primary objective is to evaluate bacterial growth and color stability between different thicknesses of 3d printed material used as a retainer .

Secondary objective is to determine the optimal thickness for use in clear aligner fabrication based on biological performance.

DETAILED DESCRIPTION:
Retainers are routinely fitted at the end of active orthodontic treatment to allow the teeth to adjust to their new positions The growing demand has led to constant improvements in materials and technologies offered by a rising number of different companies.

In recent years, major technological innovations in 3D printing, especially related to computer-aided design, biomaterials and manufacturing techniques, have enabled the production of in-office direct printed Retainers (DPRs) - representing an innovation compared to the traditional thermoformed Retainers.

Insufficient cleaning will lead to microbe's growth in retainers. The mostly found microbes are candida and staphylococcus that may include MRSA strains. Once the biofilms are formed in the retainer it's quite difficult to remove that biofilm which shows resistance to antimicrobials and difficult to clear.

orthodontic retainers hinder the sterilizing effect of saliva, which further promotes the rapid division, reproduction, and growth of colonized bacteria.

Staphylococcus aureus is most commonly found on the retainers and tends to cause bloodstream infections which can lead to serious other infections.

While several studies have assessed tooth movement, and biomechanical and clinical effects according to the design of attachments, studies investigating the thickness of the CAs are limited

ELIGIBILITY:
Inclusion Criteria:

* -Finished fixed orthodontic therapy and seeking for retention as a part of their original treatment plan.
* Good oral hygiene.
* No habits (e.g., smoking)

Exclusion Criteria:

* Medication affecting saliva.

  * intrinsic tooth discoloration.
  * Uncooperative patients.
  * Patient with periodontitis.
  * Learning difficulties and inability to read written instructions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial growth measured using colony-forming unit (CFU) count on agar plates. | from day 0 (Baseline time ) to 14 days after insertion
  Saliva samples will be collected from each participant at baseline and at day 14. Samples will be cultured on standard agar plates under aerobic conditions. After incubation, bacterial colonies will be counted, and results will be expressed in colony-forming units per milliliter (CFU/ml). A higher CFU value indicates greater bacterial growth.
  Units:
  CFU/ml
Color change of 3D printed retainers measured using spectrophotometer; ΔE calculated at day 0 and day 14. | from day 0 (baseline time ) to 14 days after insertion
  The color stability of the retainers will be assessed using a spectrophotometer (VITA Easyshade or equivalent). Color difference (ΔE) will be calculated between baseline and day 14. A ΔE > 3.3 is considered clinically perceptible. Scale range: 0-10; higher ΔE score indicates greater color change and worse color stability.
  Units:
  ΔE (Delta E) score

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mustafa Mohamed Mahmoud Dawaba Associate Professor of Orthodontics, Study Chair — Faculty of Dental Medicine, Al-Azhar University Assiut Branch; Dr. Mahmoud Mohamed Salah El-din Ibrahim Lecturer of Orthodontics, Study Chair — Faculty of Dental Medicine , Al-Azhar University Assiut Branch
Locations (1):
- Faculty of Dental Medicine , Al-Azhar University, Asyut, Egypt